CLINICAL TRIAL: NCT02512679
Title: Protocol for Related Donor Hematopoietic Stem Cell Transplantation (HSCT) for Treatment of Symptomatic Genetic Lymphohematological Diseases
Brief Title: Related Hematopoietic Stem Cell Transplantation (HSCT) for Genetic Diseases of Blood Cells
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Optimal dose obtained for engraftment and minimizing toxicity
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Lucile Packard Children's Hospital (Other)
Responsible Party: Principal Investigator, Neena Kapoor, M.D., Principal Investigator, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-06-00177
Record Dates: First submitted 2015-05-21; First posted 2015-07-31 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Stem Cell Transplantation; Bone Marrow Transplantation; Peripheral Blood Stem Cell Transplantation; Allogeneic Transplantation; Genetic Diseases; Thalassemia; Pediatrics; Diamond-Blackfan Anemia; Combined Immune Deficiency; Wiskott-Aldrich Syndrome; Chronic Granulomatous Disease; X-linked Lymphoproliferative Disease; Metabolic Diseases
Keywords: Hematopoietic Stem Cell Transplantation Pediatrics,; stem cell transplantation; bone marrow transplantation; Peripheral Blood Stem Cell Transplantation; Allogeneic Transplantation; pediatrics; Combined Immune Deficiency; Chronic Granulomatous disease
MeSH Terms: conditions — Genetic Diseases, Inborn; Thalassemia; Anemia, Diamond-Blackfan; Wiskott-Aldrich Syndrome; Granulomatous Disease, Chronic; Lymphoproliferative Disorders; Metabolic Diseases | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cyclophosphamide Dose Level 1 (Other): Cyclophosphamide given by Intravenous (IV) at a total dose of 105 mg/kg, to be divided into three doses of one 35 mg/kg dose per day, for 3 days on the first level.
  Drug to be given in combination of Busulfan, Campath and Fludarabine
  Interventions: Drug: Cyclophosphamide Dose Level 1
- Cyclophosphamide Dose Level 2 (Other): Cyclophosphamide given by intravenous (IV) at a total dose of 70 mg/kg (divided in two doses) given once a day for two days in combination with Busulfan, Campath and Fludarabine.
  Interventions: Drug: Cyclophosphamide Dose Level 2
- Cyclophosphamide Dose Level 3 (Other): Cyclophosphamide given by intravenous (IV) at total does of 35 mg/kg as a one time dose in combination with Busulfan, Fludarabine and Campath
  Interventions: Drug: Cyclophosphamide Dose Level 3
- Cyclophosphamide Dose Level 4 (Other): No cyclophosphamide given with Busulfan, Fludarabine and Campath
  Interventions: Drug: Cyclophosphamide Dose Level 4

INTERVENTIONS:
Drug: Cyclophosphamide Dose Level 1 — given by IV at a total dose of 105 mg/kg, to be divided into three doses of one 35 mg/kg dose per day, for 3 days on the first level. After ten patients the de-escalation will begin if the stopping rule is not met.
  Other Names: Cytoxan
  Arms: Cyclophosphamide Dose Level 1
Drug: Cyclophosphamide Dose Level 2 — Level 2 will be 70mg/kg in 2 divided given once a day for 2 days;
  Other Names: Cytoxan
  Arms: Cyclophosphamide Dose Level 2
Drug: Cyclophosphamide Dose Level 3 — Level 3 will be 35mg/kg as a one-time dose.
  Other Names: Cytoxan
  Arms: Cyclophosphamide Dose Level 3
Drug: Cyclophosphamide Dose Level 4 — Level 4 will be no cytoxan.
  Other Names: Cytoxan
  Arms: Cyclophosphamide Dose Level 4

SUMMARY:
Many genetic diseases of lymphohematopoietic cells (such as sickle cell anemia, thalassemia, Diamond-Blackfan anemia, Combined Immune Deficiency (CID), Wiskott-Aldrich syndrome, chronic granulomatous disease, X-linked lymphoproliferative disease, and metabolic diseases affecting hematopoiesis) are sublethal diseases caused by mutations that adversely affect the development or function of different types of blood cells. Although pathophysiologically diverse, these genetic diseases share a similar clinical course of significant progressive morbidity, overall poor quality of life, and ultimate death from complications of the disease or its palliative treatment. Supportive care for these diseases includes chronic transfusion, iron chelation, and surgery (splenectomy or cholecystectomy) for the hemoglobinopathies; prophylactic antibiotics, intravenous immunoglobulin, and immunomodulator therapies for the immune deficiencies; and enzyme replacement injections and dietary restriction for some of the metabolic diseases. The suboptimal results of such supportive care measures have led to efforts to implement more aggressive therapeutic interventions to cure these lymphohematopoietic diseases. The most logical strategies for cure of these diseases have been either replacement of the patient's own hematopoietic stem cells (HSC) with those derived from a normal donor allogeneic bone marrow transplant (BMT) or hematopoietic stem cell transplant (HSCT), or to genetically modify the patient's own stem cells to replace the defective gene (gene therapy).

DETAILED DESCRIPTION:
The present study is to evaluate de-escalation of the cyclophosphamide (CY) dose in an innovative conditioning regimen with fludarabine and alemtuzumab as additional agents to achieve immunoablation, in combination with Busulfan (BU) to achieve myeloablation. Replacement of at least part of the cyclophosphamide dose by fludarabine in the conditioning regimen would be expected to maintain immunosuppression (and, therefore, engraftment) while reducing transplant-related complications (mucositis, hepatotoxicity, cardiotoxicity, pulmonary toxicity, hemorrhagic cystitis, mucositis, and possibly GVHD), thereby improving disease-free survival rates. Similarly, the potential benefits of alemtuzumab in the proposed conditioning regimen are increased rates of hematopoietic engraftment with less toxicity than that observed with cyclophosphamide, ultimately resulting in improved immune function and enhanced quality of life (12,13). A fludarabine/alemtuzumab-based, less intensive conditioning regimen with adequate immunosuppressive activity could conceivably allow more successful engraftment of stem cells from related donors in patients with genetic lymphohematological diseases, as well as lower rates of transplant-related mortality.

Regimen-related toxicity is also believed to be a major contributing factor to GVHD (14). Therefore, conditioning regimens that cause less tissue injury may also lead to reduced GVHD. In the present study, the use of alemtuzumab in the conditioning regimen may be an added benefit, as this antibody causes T-cell depletion, thus, the risk of GVHD may also be reduced (15). The overall goal of the study is to improve the therapeutic index of HSCT by decreasing and, if possible, eliminating cyclophosphamide as a component of the pre-transplant conditioning for patients with genetic diseases of lymphohematopoiesis. The investigation will explore the risks and benefits of the proposed novel-conditioning regimen using a decreased dose of cyclophosphamide and additional immunosuppression with fludarabine and alemtuzumab to prevent graft rejection and recurrence of disease. The investigators will evaluate this regimen's impact on conditioning-related morbidity and mortality, and measure the success of the transplant procedure by engraftment and disease-free survival. If this regimen is able to successfully permit engraftment and reduce regimen-related toxicity, the next phase of treatment will test a further dose de-escalation for cyclophosphamide. It is anticipated that there will be four dose levels of cyclophosphamide in the overall study: 1) 105 mg/kg; 2) 70 mg/kg; 3) 35 mg/kg; and then finally, 4) 0 mg/kg. This study design was chosen to minimize study risks possibly associated with substitution of fludarabine and alemtuzumab for CY as immunoablation. The present protocol represents Level 1 in the study design; an amended protocol will be prepared prior to further de-escalation of the cyclophosphamide dose.

ELIGIBILITY:
Inclusion Criteria:

* All patients with lethal or sublethal genetic lymphohematological disease (such as Hemaphagocytic lymphohistiocytosis (HLH) / Familial Erythrophagocytic Lymphohistiocytosis (FEL), Hurler's Syndrome, Hunter's Syndrome, Kostmann's Syndrome, Blackfan-Diamond Anemia, Chronic granulomatous Disease (CGD), Red Cell Aplasia, CID, Sickle Cell Anemia, Thalassemia, Adreno-leukodystrophy, metachromatic leukodystrophy, Wiskott-Aldrich Syndrome, X-Linked Lymphoproliferative Disease (XLD), Metabolic diseases affecting hematopoiesis, but not limited to), who are candidates for allogeneic transplantation for their disease and have a histocompatible sibling or related donor, ages 0 to 21 years, will be candidates for this study protocol. The suitable related donor is a 10/10 or 9/10 allele Human Leukocyte Antigen (HLA) match with the patient. All patients who have previously had serious life- threatening events due to disease process may be included in the study. Patients must have adequate physical function and vital organ function to tolerate transplant procedure, as measured by:
* Cardiac: Shortening fraction >26% or left ventricular ejection fraction at rest must be > 40%.
* Hepatic: Bilirubin, Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 3x upper limit of normal (as per local laboratory) for age (with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome).
* Renal: Serum creatinine < 2x upper limit of normal for age or if serum creatinine elevated beyond normal range patient must have creatinine Clearance or Glomerular filtration rate (GFR) >50% lower limit of normal for age.
* Pulmonary: Forced expiratory volume (FEV)1, Forced Vital Capacity (FVC), and Diffusing Lung Capacity for Carbon Monoxide (DLCO) (corrected for Hgb) > 50% predicted. For patients where pulse oximetry is performed, O2 saturation > 92%
* Evaluation of iron status in patients who have received more than 12 red cell transfusions. Measurements of serum ferritin levels and MRI of the liver and heart tissue will evaluate the iron stores. If high iron load is identified in these organs further evaluation will be done to determine the suitability as transplant recipient. Should these studies indicate that chelation is necessary the following should apply: That the treating hematologist will provide the specific chelation type and timing. Evaluation of organ iron load will be part of the HSCT work-up and if high iron load is identified then the BMT team will work with the hematologist attending in developing a plan for the patient.

Exclusion Criteria:

* Karnofsky performance status < 70%, or Lansky < 40% for patients < 16 years old.
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication yet clinical symptoms progress).
* Seropositivity for the human immunodeficiency virus (HIV).
* Acute active hepatitis.
* Diagnosis of end-organ dysfunction that precludes the ability to tolerate the transplant procedure.
* Patients with a diagnosis of Fanconi Anemia are excluded.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neena Kapoor, M.D., Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: Yes
Tranplant data is reported to CIBMTR and is available to the other investigators

REFERENCES:
- [Result] Mahadeo KM, Weinberg KI, Abdel-Azim H, Miklos DB, Killen R, Kohn D, Crooks GM, Shah AJ, Kharbanda S, Agarwal R, Kapoor N. A reduced-toxicity regimen is associated with durable engraftment and clinical cure of nonmalignant genetic diseases among children undergoing blood and marrow transplantation with an HLA-matched related donor. Biol Blood Marrow Transplant. 2015 Mar;21(3):440-4. doi: 10.1016/j.bbmt.2014.11.005. Epub 2014 Nov 13. PMID 25459642
- See also: Reduced-toxicity regimen for related HSCT transplants — http://www.ncbi.nlm.nih.gov/pubmed?term=%22Biology+of+blood+and+marrow+transplantation+%3A+journal+of+the+American+Society+for+Blood+and+Marrow+Transplantation%22%5BJour%5D+AND+21%5Bvolume%5D+AND+Mahadeo%5Bauthor%5D&cmd=detailssearch

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients for bone marrow transplantation who met the eligibility criteria of diagnosis and clinical status and had histocompatible sibling donor. These patients were recruited at Children's Hospital Los Angeles and Lucille Packard Children's Hospital at Stanford University. Patients were recruited between 2006 and 2013.
Pre-assignment Details: This is a sequential dose de-escalation of Cyclophosphamide with first at 105 mg/kg total dose compared to standard 200mg/kg total dose (Arm 1). Prior to enrollment patients had to meet all eligibility criteria for allogeneic transplantation. Study closed after 1st level because all patients engrafted and none had toxicity related to transplant.
Groups:
- Cyclophosphamide Dose Level 1: Cyclophosphamide given by Intravenous (IV) at a total dose of 105 mg/kg, to be divided into three doses of one 35 mg/kg dose per day, for 3 days on the first level.
  Drug to be given in combination of Busulfan, Campath and Fludarabine
  Cyclophosphamide Dose Level 1: given by IV at a total dose of 105 mg/kg, to be divided into three doses of one 35 mg/kg dose per day, for 3 days on the first level. After ten patients the de-escalation will begin if the stopping rule is not met.
- Cyclophosphamide Dose Level 2: De-escalation of Cyclophosphamide given by Intravenous (IV) at a total dose of 70 mg/kg, to be divided into two doses of one 35 mg/kg dose per day, for 2 days
  Drug to be given in combination of Busulfan, Campath and Fludarabine
  Cyclophosphamide Dose Level 1: given by IV at a total dose of 75 mg/kg, to be divided into two doses of one 35 mg/kg dose per day, for 2 days. After ten patients the de-escalation will begin if the stopping rule is not met.
Period: Overall Study
Arm/Group | Cyclophosphamide Dose Level 1 | Cyclophosphamide Dose Level 2
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide Dose Level 1
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] — Deviation from study protocol - enrollment of 26-year-old subject with pediatric disease. Subject's data included in outcome measurements/analysis.
  years | 2.3 [.4 to 26]
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants] — Enrollment of participants was conducted in California.
  participants
    United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Neutrophil Engraftment (=/>500 Cells/uL) and Platelet Engraftment (>20K Cell/uL) at 30 Days
Description: Absolute Neutrophil Count (ANC) =/>500;(recovery of white cell count - self sustain platelet above 20,000 per cubic milimeter (20K) - evaluation by Chimerism Study (STR or FISH) at day +30
Time Frame: 30 days
Population: Subject enrolled and received Dose Level 1 of Cyclophosphamide and engrafted with Absolute Neutrophil Count (ANC) =/>500;(recovery of white cell count - self sustain platelet above 20k - evaluation by Chimerism Study (STR or FISH) at day +30.
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide Dose Level 1
Number analyzed (Participants) | 20
participants | 20

2. Primary Outcome: Number of Participants With Disease Recurrence at 1 Year Post-transplant
Description: assess rate of disease recurrence ("late relapse") due to autologous recovery of recipient hematopoiesis at one year post-HSCT.
Time Frame: 1 year
Population: All subjects who received dose level 1 of Cyclophosphamide did not experience re-occurrence of disease.
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide Dose Level 1
Number analyzed (Participants) | 20
participants | 0

3. Primary Outcome: Number of Participants Who Developed Severe Mucositis, Veno-occlusive Disease (VOD), Toxicity of the Kidney, Liver, or Gastrointestinal (GI) Tract up to 1 Year Post-transplant
Description: Assessment of conditioning regimen related toxicity was evaluated and documented with daily assessment during hospitalization and post-transplant follow-up up to one year. None of the subjects developed VOD necessitating any therapeutic intervention, severe mucositis, or toxicity of the Kidney, Liver or Gastrointestinal.
Time Frame: 1 year
Population: Subjects who received dose level 1 of Cyclophosphamide did not experience veno-occlusive disease, organ failure or severe mucositis.
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide Dose Level 1
Number analyzed (Participants) | 20
participants
  Veno-Occlusive Disease | 0
  Viral Infection | 8
  Toxicity of Kidney, Liver, or Gastrointestinal | 0
  Severe Mucositis | 0

4. Secondary Outcome: Number of Participants Who Developed Graft-Versus-Host-Disease (GVHD) as Determined by the Glucksberg Scale
Description: Clinical evaluation on a daily basis during hospitalization and at each post transplant clinical visit, up to one year, to determine incidence of acute and chronic graft-versus-host disease using Glucksberg grading scale. Acute graft-versus-host disease (aGVHD) develops within the first three months after transplantation and appears as a skin rash, often accompanied by hyperbilirubenemia, abnormal liver enzymes and gastrointestinal symptoms, as diarrhea, nausea and vomiting. Level of aGVHD is graded from 1-4. Chronic GVHD, typically a late complication of Blood and Marrow Transplantation (BMT) characterized by skin changes, sometimes sclerotic changes, with joint contractures, liver function abnormality, gastrointestinal symptoms and sometime other organ involvement such as eyes, lungs, and obliterative bronchiolitis (OB). Chronic GVHD is graded as absent, limited, or extensive.
Time Frame: 1 yr
Population: Subjects who received dose level 1 of Cyclophosphamide were revaluated for graft-versus-host disease (GVHD) post transplantation.
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide Dose Level 1
Number analyzed (Participants) | 20
participants
  Acute GVHD (Grade 1-2) | 10
  Acute GVHD (Grade 3-4) | 0
  Chronic GVHD | 0

5. Secondary Outcome: Number of Participants Who Were Disease Progression-Free and Death-Free at 1 Year Post-transplant
Description: Evaluation for engraftment, correction of the disease, transplant related complications and event-free survival and overall survival of the subjects post-transplant was undertaken by standard measures and evaluation of disease with disease-specific testing.
Time Frame: 1 yr
Population: Subjects receiving dose level 1 of Cyclophosphamide event free survival post transplant at 100 days was 95% and 90% 1 year.
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide Dose Level 1
Number analyzed (Participants) | 20
participants
  100 Day Event Free Survival Post Transplant | 19
  One Year Event Free Survival Post Transplant | 18
  Disease Progression-Free | 20

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the course of the study up to 2 years post transplantation. Subjects were evaluated for post transplant complications related to conditioning, such as VOD, GVHD, infections and engraftment failure.
Arm/Group | Cyclophosphamide Dose Level 1
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide Dose Level 1 (N=20)
Death due to pre-exisiting mucormycosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject had pretransplant history of mucormycosis infection. Patient was received anti-fungal medications.
Death due to interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject developed interstitial pneumonia on Day +187 post transplant. Onset thought to be community acquired pneumonia.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide Dose Level 1 (N=20)
Cytomegalovirus (CMV) infection (Blood and lymphatic system disorders) | 5 (5) — Re-activation of cytomegalovirus (CMV) in 5/20 enrolled subjects documented by blood CMV Polymerase Chain Reaction (PCR) test.
Epstein-Barr Virus (EBV) (Blood and lymphatic system disorders) | 1 (1) — Epstein-Barr Virus (EBV) was documented to be positive in 1/20 subjects enrolled in the study; confirmed by Polymerase Chain Reaction (PCR).
Adenovirus (Blood and lymphatic system disorders) | 1 (1) — Adenovirus was detected in one (1) enrolled subject by blood PCR.

LIMITATIONS AND CAVEATS:
De-escalation was not ensued. All enrolled subjects engrafted without toxicity for dose level one.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No